CLINICAL TRIAL: NCT03360214
Title: A Comparison of Pulsed Electromagnetic Fields (PEMF) and Pectoral (PEC) Interfascial Blocks on Postoperative Pain Reduction in Patients Undergoing Mastectomy and Tissue Expander Reconstruction
Brief Title: PEMF and PEC Blocks in Mastectomy Reconstruction Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Christine Hsu Rohde, MD, Professor of Plastic and Reconstructive Surgery, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAQ4708
Record Dates: First submitted 2017-11-27; First posted 2017-12-04 (Actual); Results first posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Female
Keywords: Mastectomy; Tissue expander; PEMF; PIB
MeSH Terms: interventions — Bupivacaine; Sodium Chloride; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Active PEMF + Treatment PIB (Other): Participants will receive an active device (Pulsed Electromagnetic Field (PEMF) Device) and active drug (Bupivacaine Hydrochloride or Ropivacaine HCl).
  Interventions: Drug: Bupivacaine Hydrochloride; Device: Pulsed Electromagnetic Field (PEMF) Device; Drug: Ropivacaine Hydrochloride
- Active PEMF + Sham PIB (Other): Participants will receive an active device (Pulsed Electromagnetic Field (PEMF) Device) and placebo drug.
  Interventions: Other: Placebo Drug; Device: Pulsed Electromagnetic Field (PEMF) Device
- Sham PEMF + Treatment PIB (Other): Participants will receive a placebo device and active drug (Bupivacaine Hydrochloride or Ropivacaine HCl).
  Interventions: Drug: Bupivacaine Hydrochloride; Other: Placebo Device; Drug: Ropivacaine Hydrochloride
- Sham PEMF + Sham PIB (Other): Participants will receive placebo drug and placebo device.
  Interventions: Other: Placebo Drug; Other: Placebo Device

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — For active drug, 0.25% marcaine, will be used.
  Other Names: Marcaine; PIB
  Arms: Active PEMF + Treatment PIB; Sham PEMF + Treatment PIB
Other: Placebo Drug — For sham drug, 0.9% saline, will be used.
  Other Names: Saline
  Arms: Active PEMF + Sham PIB; Sham PEMF + Sham PIB
Device: Pulsed Electromagnetic Field (PEMF) Device — The pulsed electromagnetic field signal will consist of a 2-m sec burst of 27.12 megahertz (MHz) radiofrequency sinusoidal waves repeating at 2 bursts/second.
  Other Names: Sofpulse; Torino II
  Arms: Active PEMF + Sham PIB; Active PEMF + Treatment PIB
Other: Placebo Device — Sham devices will appear identical to and will be used in exactly the same manner as active devices but will produce no electromagnetic field.
  Arms: Sham PEMF + Sham PIB; Sham PEMF + Treatment PIB
Drug: Ropivacaine Hydrochloride — For active drug, 0.25% naropin, will be used.
  Other Names: Naropin; PIB
  Arms: Active PEMF + Treatment PIB; Sham PEMF + Treatment PIB

SUMMARY:
This is a prospective randomized controlled double-blind interventional study comparing the effect of pulsed-electromagnetic field device (PEMF), pectoral interfascial block (PIB), and placebo on postoperative pain control. This study has the interdisciplinary cooperation of the regional anesthesia group, and the breast and plastic surgery divisions. All female patients with breast cancer evaluated at Columbia University Medical Center (CUMC) who are undergoing unilateral or bilateral mastectomy with tissue expander reconstruction will be offered enrollment in this prospective study.

DETAILED DESCRIPTION:
Chronic pain after mastectomy, or breast tissue removal, is very common with almost half of women experiencing some type of residual pain and even 13% characterizing it as severe. Poor acute postoperative pain control is not only associated with development of chronic pain, but has also been shown to be associated with delayed wound healing. Therefore, optimization of postoperative pain control is paramount not just for patient comfort, but to decrease immediate and long-term postoperative complications.

There are two adjunctive modes of perioperative pain control currently in use at Columbia University Medical Center (CUMC). The first mode uses pulsed electromagnetic fields (PEMF) and consists of a noninvasive device placed over dressings around the surgical site. The second is a regional anesthetic and -the pectoral interfascial block (PIB) in which a long-lasting local anesthetic (bupivacaine/ropivacaine) is injected into the surgical dissection area. Both of these techniques for postoperative analgesia have been shown to be effective in different types of breast surgery, but there is no current literature comparing the two modalities in their efficacy in reducing postoperative pain. There is also no current literature in their efficacy in the mastectomy and tissue expander patient population. The proposed trial is a prospective, randomized, controlled, double-blind trial to evaluate the efficacy of these two modalities of postoperative analgesia in patients undergoing mastectomy and tissue expander reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be female
* Subjects must be 18 years or older
* Subjects must be undergoing unilateral or bilateral mastectomy with tissue expander reconstruction

Exclusion Criteria:

* Allergy to all narcotic medications
* Intake of any chronic opioids or pain medications preoperatively for a chronic condition or chronic use.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Rohde, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham PEMF + Treatment PIB: Participants will receive a placebo device and active drug (Bupivacaine Hydrochloride).
  Bupivacaine Hydrochloride: For active drug, 0.25% marcaine, will be used.
  Placebo Device: Sham devices will appear identical to and will be used in exactly the same manner as active devices but will produce no electromagnetic field.
Period: Overall Study
Arm/Group | Active PEMF + Treatment PIB | Active PEMF + Sham PIB | Sham PEMF + Treatment PIB | Sham PEMF + Sham PIB
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active PEMF + Treatment PIB: Participants will receive an active device (Pulsed Electromagnetic Field (PEMF) Device) and active drug: 0.25% Bupivacaine Hydrochloride or 0.25% Ropivacaine HCl.
- Active PEMF + Sham PIB: Participants will receive an active device (Pulsed Electromagnetic Field (PEMF) Device) and placebo drug: 0.9% saline.
- Sham PEMF + Treatment PIB: Participants will receive a placebo device (identical appearance to active device, but produces no electromagnetic field) and active drug: 0.25% Bupivacaine Hydrochloride.
- Total: Total of all reporting groups
Arm/Group | Active PEMF + Treatment PIB | Active PEMF + Sham PIB | Sham PEMF + Treatment PIB | Sham PEMF + Sham PIB | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Continuous [Median (Full Range); unit: years] | 50 [32 to 68] | 53 [31 to 64] | 48 [33 to 69] | 53 [36 to 60] | 50 [31 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 15 | 15 | 60
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 5 | 7 | 23
  Not Hispanic or Latino | 10 | 9 | 10 | 8 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 3 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 4 | 6 | 18
  White | 9 | 10 | 8 | 4 | 31
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 15 | 15

OUTCOME MEASURES:

1. Primary Outcome: Score on Visual Analog Scale (VAS) - 1 Hour Post-intervention
Description: Pain level will be measured using the VAS scale. Subjects will rate their pain level on a scale of 0-10. Number "0" indicates no pain and number "10" indicates terrible pain.
Time Frame: 1 hour post-intervention
Population: 4 participants declined to do the VAS assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active PEMF + Treatment PIB | Active PEMF + Sham PIB | Sham PEMF + Treatment PIB | Sham PEMF + Sham PIB
Number analyzed (Participants) | 14 | 15 | 13 | 14
score on a scale | 6.64 (2.76) | 6.67 (2.29) | 4.62 (3.57) | 6.93 (2.4)

2. Secondary Outcome: Quality of Recovery Questionnaires (QoR) - 1 Hour Post-intervention
Description: Quality of recovery will be measured using QoR. QoR is a 15-item self-reported questionnaire, with each response on a scale of 0-10 pertaining to patient's comfort, support system, pain, well being, and ability to carry out daily activities. The total score range is 0 to 150, with a higher score indicating a better quality of recovery.
Time Frame: 1 hour post-intervention
Population: Some participants in each arm declined to do the QoR assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active PEMF + Treatment PIB | Active PEMF + Sham PIB | Sham PEMF + Treatment PIB | Sham PEMF + Sham PIB
Number analyzed (Participants) | 8 | 10 | 11 | 12
score on a scale | 82.88 (25.67) | 90.90 (36.14) | 82.91 (35.24) | 77.50 (16.84)

3. Secondary Outcome: Quality of Recovery Questionnaires (QoR) - 3 Weeks Post-intervention
Description: as for outcome 2
Time Frame: 3 weeks post-intervention
Population: 1 participant declined to do the QoR assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active PEMF + Treatment PIB | Active PEMF + Sham PIB | Sham PEMF + Treatment PIB | Sham PEMF + Sham PIB
Number analyzed (Participants) | 15 | 15 | 15 | 14
score on a scale | 122 (23.79) | 123.27 (18.77) | 125.93 (20.29) | 121 (26.92)

4. Primary Outcome: Score on Visual Analog Scale (VAS) - 3 Weeks Post-intervention
Description: as for outcome 1
Time Frame: 3 weeks post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active PEMF + Treatment PIB | Active PEMF + Sham PIB | Sham PEMF + Treatment PIB | Sham PEMF + Sham PIB
Number analyzed (Participants) | 15 | 15 | 15 | 15
score on a scale | 2.53 (2.07) | 2.00 (2.20) | 2.00 (1.89) | 2.67 (2.89)

ADVERSE EVENTS:
Time Frame: Up to 3 weeks
Groups:
- Active PEMF + Bupivacaine Hydrochloride: Participants will receive an active device (Pulsed Electromagnetic Field (PEMF) Device) and active drug: 0.25% Bupivacaine Hydrochloride.
- Active PEMF + Ropivacaine HCl: Participants will receive an active device (Pulsed Electromagnetic Field (PEMF) Device) and active drug: 0.25% Ropivacaine HCl.
- Active PEMF + Placebo: Participants will receive an active device (Pulsed Electromagnetic Field (PEMF) Device) and placebo drug: 0.9% saline.
- Sham PEMF + Bupivacaine Hydrochloride: Participants will receive a placebo device (identical appearance to active device, but produces no electromagnetic field) and active drug: 0.25% Bupivacaine Hydrochloride.
- Sham PEMF + Placebo: Participants will receive placebo drug and placebo device.
Arm/Group | Active PEMF + Bupivacaine Hydrochloride | Active PEMF + Ropivacaine HCl | Active PEMF + Placebo | Sham PEMF + Bupivacaine Hydrochloride | Sham PEMF + Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/1 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/1 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/14 | 0/1 | 0/15 | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Due to drug shortage, Ropivacaine was used in place of Bupivacaine in 1 participant. Bupivacaine and Ropivacaine are FDA-approved local anesthetics currently used in pectoral interfascial blocks for breast surgery patients. Bupivacaine and Ropivacaine are both long-acting local anesthetics with a similar mechanism of action.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/14/NCT03360214/Prot_SAP_000.pdf